CLINICAL TRIAL: NCT04264429
Title: Effect of the Infrapatellar Strap and Elastic Band on the Pain, Agility, Balance and Lower Limb Function Athletes With Patellofemoral Pain Syndrome
Brief Title: Effect of the Infrapatellar Strap and Elastic Band Iin Athletes With Patellofemoral Pain Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Christiane Macedo, Principal investigator and Professor., Universidade Estadual de Londrina
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Strap in patelofemoral pain.
Record Dates: First submitted 2019-12-02; First posted 2020-02-11 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Recruitment
Keywords: Patellofemoral Pain Syndrome; Physiotherapy; Knee; Orthoses
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Compression Bandages

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Infrapatellar strap (Experimental): This group will perform the functional tests with the infrapatellar strap positioned on the painful knee.
  Interventions: Device: Infrapatellar strap
- Elastic Band (Experimental): This group will perform the functional tests with the elastic band positioned on the painful knee.
  Interventions: Other: Elastic band
- Control (No Intervention): This group will perform the functional tests without elastic band or infrapatellar strap positioned on the painful knee.

INTERVENTIONS:
Device: Infrapatellar strap — Orthotic device which is positioned over the patellar tendon
  Other Names: Infrapatellar strip
  Arms: Infrapatellar strap
Other: Elastic band — Orthotic device which is positioned over the patellar tendon
  Other Names: Elastic bandage
  Arms: Elastic Band

SUMMARY:
Patellofemoral Pain Syndrome (PPS) is common in athletes, especially when performing jumps. To reduce pain and improve functionality, orthoses such as the infrapatellar strip (IPS) and functional bandage (FB) are indicated, but their effects are controversial. The objective is to evaluate the effect of IPS and FB on lower limb pain, agility, balance and strength in athletes with PPS. Will be evaluated 25 athletes with PPS (10 women and 15 men), who will answer the sample characterization questionnaires, pain scale and performed the Side Hope Test (SHT), modified star excursion balance test (SEBTm) and Sit to Stand 30 in seconds (STS30 ") to analyze lower limb agility, balance and strength, respectively. Three repetitions of each functional test will be performed, with an interval of one minute between repetitions and tests. Still, the tests will be developed with IPS, with FB and without any orthosis, with previously randomized sequence. Expected to establish the effects of IPS and FB for athletes with PPS.

DETAILED DESCRIPTION:
The research was approved by the ethics committee of the institution. The sample size was calculated in 18 athletes, but when considering losses 25 athletes (10 women and 15 men) were recruited.

Athletes will be over 18 years old, from different sports or teams, with a minimum of six hours / week of training / competition, with complaints of anterior knee pain (DAJ) greater than 3 on the visual analog scale (VAS), rating lower than or equal to 82 (tendency to patellofemoral disorder) in the Anterior Knee Pain Scale (AKPS) and score lower than or equal to 83 (fair or poor) on the Lysholm questionnaire. Exclusion criteria will be the history of other lower limb injuries or surgery; diabetes or altered sensitivity in the plantar region; medication and physical therapy use in the last three months.

For data collection athletes will answer the sample characterization questionnaires, AKPS and Lysholm.

Modified star excursion balance test (SEBTm), Side Hope test (SHT) and 30 second sit-up test (SL30 '') will be applied, at random and with prior familiarization, for the analysis of dynamic balance, agility and lower limb strength, respectively.

It will also be randomized the tests with Infrapatellar Strap, Elastic Bandage and without orthosis (control), developed in three different days with 96 hours interval. To apply the infrapatellar strap and elastic bandage, the athlete was positioned standing with slight knee flexion, with heel support on a pre-established surface (relaxed patellar tendon). The Infrapatellar Strap and Elastic Bandage will be positioned over the patellar tendon, with moderate pressure, on the lower limb complaining of pain.

The tests: SEBTm test, Side Hope test (SHT), and 30-second sit-up (STS 30 '') will be repeated three times, with a one-minute interval between trials and five minutes between tests. At the beginning and end of each test, the analogue visual pain scale (VAS) for knee pain will be applied.

Statistical data will be analyzed using the Statistical Package of Social Science (SPSS®) program, version 22 and a significance level of 5% (p <0.05). ANOVA two way test will be used to compare groups, times and their interaction.

ELIGIBILITY:
Inclusion Criteria:

* Athletes will be over 18 years old,
* From different sports or teams,
* With a minimum of six hours / week of training / competition,
* With complaints of anterior knee pain (DAJ) greater than 3 on the visual analog scale (VAS)
* Rating lower than or equal to 82 (tendency to patellofemoral disorder) in the Anterior Knee Pain Scale (AKPS)
* Score lower than or equal to 83 (fair or poor) on the Lysholm questionnaire.

Exclusion Criteria:

* History of other lower limb injuries or surgery,
* Diabetes,
* Altered sensitivity in the plantar region,
* Medication to pain,
* Physical therapy use in the last three months.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-03-05 (Estimated); Primary Completion 2020-05-05 (Estimated); Study Completion 2020-10-05 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity | Evaluations will be conducted throughout the project data collection. The evaluations have an average time of three months.
  The pain will be evaluated before and after the functional tests with infrapatellar strap and elastic band, through the analogue visual pain scale (with pain characterization from zero to ten).
Balance - Modified star excursion balance test (SEBTm) | Evaluations will be conducted throughout the project data collection. The evaluations have an average time of three months.
  For the analysis of SEBTm the normalization of the directions will be develop througt the length ot the lower limb of each participant (maximum distance reached in 3 directions (anteior, postero-lateral and postero-medial) / (limb length x 3) x 100 = percentage of the three directions. Distance traveled in centimeters (on a measuring tape) in the anterior, postero-medial and postero-lateral directions.
Agility - Side Hope test (SHT) | Evaluations will be conducted throughout the project data collection. The evaluations have an average time of three months.
  For the SHT analysis will be consideres the time requered for the athlete to perform 10 lateral jumps was considered.
Endurance - 30 second sit to stand test (STS30 '') | Evaluations will be conducted throughout the project data collection. The evaluations have an average time of three months.
  For the 30" Sit and Lift Test it will be considered for analysis only complete cycles with full knee extension and seat weight unloading.

CONTACTS AND LOCATIONS:
Overall Officials: Christiane S Macedo, Principal Investigator — State University of Londrina
Locations (1):
- University Hospital of the State University of Londrina, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coburn SL, Barton CJ, Filbay SR, Hart HF, Rathleff MS, Crossley KM. Quality of life in individuals with patellofemoral pain: A systematic review including meta-analysis. Phys Ther Sport. 2018 Sep;33:96-108. doi: 10.1016/j.ptsp.2018.06.006. Epub 2018 Jun 28. PMID 30059951
- [Background] Straub RK, Cipriani DJ. Influence of infrapatellar and suprapatellar straps on quadriceps muscle activity and onset timing during the body-weight squat. J Strength Cond Res. 2012 Jul;26(7):1827-37. doi: 10.1519/JSC.0b013e318234e81d. PMID 21912298
- [Background] Collins NJ, Barton CJ, van Middelkoop M, Callaghan MJ, Rathleff MS, Vicenzino BT, Davis IS, Powers CM, Macri EM, Hart HF, de Oliveira Silva D, Crossley KM. 2018 Consensus statement on exercise therapy and physical interventions (orthoses, taping and manual therapy) to treat patellofemoral pain: recommendations from the 5th International Patellofemoral Pain Research Retreat, Gold Coast, Australia, 2017. Br J Sports Med. 2018 Sep;52(18):1170-1178. doi: 10.1136/bjsports-2018-099397. Epub 2018 Jun 20. PMID 29925502
- [Background] de Vries A, Zwerver J, Diercks R, Tak I, van Berkel S, van Cingel R, van der Worp H, van den Akker-Scheek I. Effect of patellar strap and sports tape on pain in patellar tendinopathy: A randomized controlled trial. Scand J Med Sci Sports. 2016 Oct;26(10):1217-24. doi: 10.1111/sms.12556. Epub 2015 Sep 17. PMID 26376953